CLINICAL TRIAL: NCT01760174
Title: A Randomized Double Blind Trial Comparing the Effect of Transversus Abdominal Plane-catheter and Epidural Catheter on Postoperative Pain After Open Gynecologic Surgery
Brief Title: Comparing the Effect of TAP-catheter and Epidural Catheter on Postoperative Pain After Open Gynecologic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of logistic and practical reasons.
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Nils Bjerregaard, Consultant Anesthetist, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-20120041
Record Dates: First submitted 2012-07-26; First posted 2013-01-04 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Pain, Postoperative
Keywords: Transversus abdominis plane catheter
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacain-infusion in epidural catheter (Active Comparator): Bupivacain-infusion in epidural catheter and intermittent isotonic potassium chloride bolus in transversus abdominis plane catheter.
  Interventions: Drug: Bupivacain-infusion in epidural catheter
- Ropivacaine bolus in transversus abdominis plane catheter (Active Comparator): Intermittent ropivacaine bolus in bilateral transversus abdominis plane catheter and isotonic potassium chloride infusion in epidural catheter.
  Interventions: Drug: Ropivacaine bolus in transversus abdominis plane catheter

INTERVENTIONS:
Drug: Ropivacaine bolus in transversus abdominis plane catheter — Ropivacaine 7,5 mg/ml, 10-25 ml in each catheter, depending on patient weight, the total dose of ropivacaine is kept less than 3 mg/kg for every bolus. Bolus is given every 6 hours, the first bolus is given just after induction of general anesthesia and the last bolus after 24 hours.
  In the epidural catheter a bolus of 8 ml isotonic potassium chloride is given and an infusion of isotonic potassium chloride, 4-7 ml/t depending on patient height is started and runs for the first 24 hours.
  Arms: Ropivacaine bolus in transversus abdominis plane catheter
Drug: Bupivacain-infusion in epidural catheter — Isotonic potassium chloride, 10-25 ml in each transversus abdominis catheter, depending on patient weight. Bolus is given every 6 hours, the first bolus is given just after induction of general anesthesia and the last bolus after 24 hours.
  In the epidural catheter a bolus of 8 ml bupivacaine 2,5 mg/ml is given and an infusion of isotonic potassium chloride, 4-7 ml/t depending on patient height is started and runs for the first 24 hours
  Arms: Bupivacain-infusion in epidural catheter

SUMMARY:
This study compares the effect on postoperative pain of bolus administration of ropivacaine in Transversus abdominis plane catheter and continuous bupivacain-infusion in epidural catheters following open gynecologic surgery.The study is double blind. The hypothesis is that the effect of the two modes of pain treatment are equal.

DETAILED DESCRIPTION:
Patients for open gynecologic surgery will all receive both an epidural catheter and bilateral transversus abdominis plane (:TAP) catheters. After randomization in to two groups the patients receive either 1) intermittent boluses of ropivacaine in the TAP-catheters and isotonic potassium chloride-infusion i the epidural catheters or 2) intermittent isotonic potassium chloride-boluses i the TAP-catheters and bupivacain-infusion in the epidural catheters.

The investigators record pain-score and consumption of opioids in the first 24 hours postoperatively as well as thermoanalgesia at dermatome-levels th10-th12.

The investigators assume that the effect on postoperative pain after open gynecologic surgery is equal in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for open gynecologic surgery
* acceptance to participate

Exclusion Criteria:

* allergies to local analgetics
* daily use of strong opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Pain-score on numerical rating scale | 4 hours after first bolus in tranversus abdominis catheters

SECONDARY OUTCOMES:
Administration of opioids | The first 24 hours after surgery.
Pain-score on numerical rating scale | 8 hours after first bolus in tranversus abdominis catheters
Pain-score on numerical rating scale | 24 hours after first bolus in tranversus abdominis catheters

OTHER OUTCOMES:
Thermoanalgesia at dermatome-level th10-th12 | 4 hours after first bolus in TAP-catherter

CONTACTS AND LOCATIONS:
Overall Officials: Nils F Bjerregaard, M.D., Principal Investigator — Aalborg University Hospital; Bodil S Rasmussen, M.D. + PhD, Study Director — Aalborg Sygehus; Lone Nikolajsen, M.D, PhD, Study Chair — Aarhus University Hospital; Thomas F Bendtsen, MD, PhD, Study Chair — Aarhus University Hospital
Locations (1):
- Aalborg Hospital, Aalborg, Region Nord, Denmark